CLINICAL TRIAL: NCT07106840
Title: Identification of Autism Traits in Adolescents With Social Anxiety Disorder and Evaluation of Their Association With the Broader Autism Phenotype in Their Parents
Brief Title: Autism Traits in Adolescents With Social Anxiety Disorder: Associations With Parental Broader Autism Phenotype
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Şermin Bilgen Ulgar, Child and Adolescent Psychiatry Specialist, Ankara City Hospital Bilkent
Other Study IDs: AnkaraCH_SAD_Autism_2025_01; E2-24-6099 (Other: Ankara Bilkent City Hospital Ethics Committee)
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Social Anxiety Disorder (SAD); Autistic Disorder
Keywords: Phobia, Social; Anxiety; Autistic Disorder; Parents; Social Interaction
MeSH Terms: conditions — Phobia, Social; Autistic Disorder; Anxiety Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational study with no intervention applied.

SUMMARY:
This observational study aims to examine autism-related traits in adolescents diagnosed with social anxiety disorder (SAD) and to evaluate their associations with broader autism phenotype (BAP) features in their parents. A total of 109 adolescents aged 11-17 and their parents were included. Standardized scales were used to assess social anxiety severity and autism traits in adolescents, and BAP characteristics in parents.

DETAILED DESCRIPTION:
Autism spectrum traits and social anxiety share clinical and cognitive features, particularly in the domains of social communication and interaction. These overlaps suggest that autistic traits may be present in adolescents diagnosed with social anxiety disorder (SAD), even in the absence of a formal autism diagnosis. Furthermore, the concept of the broader autism phenotype (BAP) suggests that subclinical autism-related features may be observed in parents of individuals with autism traits.

This study includes 109 adolescents (aged 11-17) diagnosed with SAD and their parents. The adolescents completed a standardized scale assessing social anxiety severity, while parents completed the Social Responsiveness Scale (SRS) for their children and the Autism Spectrum Quotient (AQ) to assess BAP characteristics in themselves. The study aimed to explore the associations between adolescents' autism-related traits and their social anxiety severity, and to evaluate how parental BAP scores (particularly fathers') may be associated with these traits.

Note: This study involved prospective recruitment and data collection; however, registration was completed retrospectively after the study was completed.

ELIGIBILITY:
Inclusion Criteria:

Adolescents aged 11-17 years diagnosed with Social Anxiety Disorder (SAB). Availability of at least one biological parent willing to participate. Ability to provide informed consent/assent.

Exclusion Criteria:

Presence of intellectual disability or severe neurological disorder. Comorbid psychiatric diagnoses that could interfere with assessment (e.g., psychosis).

Non-fluency in the language of assessment.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study included 109 adolescents aged 11-17 years diagnosed with Social Anxiety Disorder, along with their biological parents. The sample consisted of 87 females and 22 males. Participants were recruited prospectively from clinical outpatient settings.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Social Anxiety Severity | At baseline
  Severity of social anxiety symptoms measured by the Social Anxiety Disorder Severity Scale - Child Form.

SECONDARY OUTCOMES:
Autism Traits in Adolescents | At baseline
  Autism spectrum traits in adolescents assessed by the Social Responsiveness Scale, completed by parents.

OTHER OUTCOMES:
Parental Broader Autism Phenotype | At baseline
  Parental broader autism phenotype evaluated using the Autism Spectrum Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Şermin Bilgen Ulgar, Medical Doctor, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon reasonable request with qualified researchers, in accordance with ethical approvals and participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF